CLINICAL TRIAL: NCT02562898
Title: A Study of the Safety, Immunopharmacodynamics and Anti-tumor Activity of Ibrutinib Combined With Gemcitabine and Nab-Paclitaxel in Patients With Metastatic Pancreatic Adenocarcinoma
Brief Title: Ibrutinib Combined With Gemcitabine and Nab-Paclitaxel in Patients With Metastatic Pancreatic Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Margaret Tempero (Other)
Collaborators: Stand Up To Cancer (Other); Lustgarten Foundation (Other)
Responsible Party: Sponsor-Investigator, Margaret Tempero, Professor, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 144525; NCI-2015-01780 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2015-09-03; First posted 2015-09-29 (Estimated); Results first posted 2020-07-16 (Actual); Last update posted 2021-05-06 (Actual); Status verified 2021-04

CONDITIONS: Metastatic Pancreatic Adenocarcinoma
MeSH Terms: interventions — ibrutinib; Paclitaxel; Albumin-Bound Paclitaxel; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dose escalation for safety and toxicity (Experimental): All patients in phase Ib dosing escalation with extended safety and toxicity cohorts will start treatment with daily dosing of ibrutinib concurrently with standard doses of gemcitabine and nab-paclitaxel. Ibrutinib (560 mg/day, 840 mg/day, or 420 and 280 mg/day if de-escalation is necessary) will be started on day 1. Approximately patients 15-30 will be enrolled in escalation and extended safety cohort.
  Interventions: Drug: Ibrutinib; Drug: Paclitaxel; Drug: Gemcitabine
- Immune Response cohort (Experimental): Subjects who are assigned to the Immune Response Cohort will have a biopsy before starting ibrutinib-only therapy. They will then receive ibrutinib for 7 days and have a second biopsy after completing the ibrutinib-only therapy, before starting the combination of chemotherapy with ibrutinib. Approximately 20 patients will be enrolled in this arm.
  Interventions: Drug: Ibrutinib; Drug: Paclitaxel; Drug: Gemcitabine

INTERVENTIONS:
Drug: Ibrutinib — 560, 840, 420, or 280mg, orally once per day - 4 week cycle
  Other Names: PCI-32765
Drug: Paclitaxel — 125mg/m2 IV Day 1, 8, and 15 - 4 week cycle
  Other Names: Abraxane, Taxol
Drug: Gemcitabine — 1000mg/m2 IV Day 1, 8, and 15 - 4 week cycle
  Other Names: Gemzar

SUMMARY:
Gemcitabine and nab-paclitaxel is a standard regimen (NCCN, Category 1) for patients with metastatic pancreatic ductal adenocarcinoma (PDAC). However, further improvement in treatment is needed. Increasingly, the nature of the immune infiltrate in PDAC appears to be tumor promoting. In preclinical studies, ibrutinib treatment, presumably by reprogramming B cells, results in increased CD8+ T cells to assist in tumor control. Preclinical studies of ibrutinib plus gemcitabine show superior antitumor effects compared to gemcitabine alone in both orthotopic murine pancreatic cancer cell line grafts and in genetically engineered mouse models. Thus, the investigators propose a clinical trial of ibrutinib plus the standard gemcitabine based regimen of gemcitabine and nab-paclitaxel, evaluating safety, then efficacy and including correlative studies.

DETAILED DESCRIPTION:
Pancreatic adenocarcinoma (PDAC) represents the fourth leading cause of cancer-related mortality in the United States, with an estimated 39,950 deaths attributable to PDAC in 2014 (http://seer.cancer.gov/statfacts/html/pancreas.html). Over 90% of patients have inoperable disease at presentation, at which point systemic therapy becomes the primary form of treatment.

Treating PDAC has been challenging and few approved drugs are available. Recently, however, some breakthroughs have occurred, raising hope that this aggressive disease can be better controlled. FOLFIRINOX, a combination of 5FU, oxaliplatin, and irinotecan, has been found to be substantially superior to treatment of gemcitabine alone in patients with metastatic disease and good performance status. Similarly, gemcitabine and nab-paclitaxel, a regimen with less non-hematologic toxicity, demonstrated improved overall survival and progression-free survival compared to gemcitabine alone. Both of these combinations or modifications of these combinations are now front line options for patients with good performance status. Furthermore, these improvements in survival, however incremental, now afford patients with pancreatic cancer time to participate in and possibly benefit from clinical trials of novel therapeutics.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed metastatic pancreatic adenocarcinoma
* Stage IV disease (measurable disease NOT required)
* Intact primary tumor
* CA19-9 greater than 75 units
* Eastern Cooperative Oncology Group (ECOG) performance score of 0-1
* At least 18 years of age
* Female patients who are not of child-bearing potential, and fertile female patients of child-bearing potential, who agree to use adequate contraceptive measures, who are not breastfeeding, and who have a negative serum or urine pregnancy test within 72 hours prior to start of randomization.
* Fertile male patients willing to use adequate contraceptive measures.
* Adequate bone marrow function:

  * Absolute neutrophil count (ANC) ≥ 1500/microliter (uL)
  * platelet count ≥ 100,000/uL
  * hemoglobin ≥ 9.0 g/dL
* Adequate hepatic function:

  * Total bilirubin ≤ 1.5 X ULN (unless bilirubin rise due to Gilbert's syndrome)
* Aspartate amino transferase (AST) (SGOT) ≤ 3.0 X ULN; ≤5.0X ULN if liver metastases are present.
* Alanine aminotransferase (ALT) (SGPT) ≤ 3.0 X ULN; ≤0 5.0X ULN if liver metastases are present.
* Adequate renal function (defined as serum creatinine ≤ 1.5 X ULN)
* Ability to understand the nature of this study protocol, comply with study and/or follow-up procedures, and give written informed consent
* Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests, and other study procedures.

Exclusion Criteria:

* Any prior systemic or investigational therapy for metastatic pancreatic cancer. Systemic therapy administered alone or in combination with radiation in the adjuvant or neoadjuvant setting is permissible as long as it was completed > 6 months prior to the time of study registration.
* History of other diseases, metabolic dysfunction, physical examination findings, or clinical laboratory findings giving reasonable suspicion of a disease or condition that, in the opinion of the investigator, renders the subject at high risk from treatment complications or might affect the interpretation of the results of the study.
* History of previous malignancy (except basal cell) within 5 years.
* Life expectancy of <3 months.
* Inability to undergo two sequential Endoscopic Ultrasound (EUS)-directed core biopsies of the primary tumor.
* Presence of known central nervous system or brain metastases.
* Known human immunodeficiency virus (HIV) infection.
* History of stroke or intracranial hemorrhage within 6 months prior to enrollment.
* Known bleeding disorders (e.g., von Willebrand's disease or hemophilia).
* Patients receiving warfarin or other Vitamin K antagonists. However, if therapeutic anticoagulation is necessary, low molecular weight heparin (LMWH) is the anticoagulant of choice.
* Currently active, clinically significant cardiovascular disease, such as uncontrolled arrhythmia or Class 3 or 4 congestive heart failure as defined by the New York Heart Association Functional Classification; or a history of myocardial infarction, unstable angina, or acute coronary syndrome within 6 months prior to randomization.
* Current peripheral sensory neuropathy > Grade 1
* Major surgery within 4 weeks of the start of study treatment (defined as those surgeries that require general anesthesia. Insertion of a vascular access device is NOT considered major surgery.
* Requires treatment with a strong cytochrome P450 (CYP) 3A inhibitor.
* Unable to swallow capsules or has malabsorption syndrome, disease significantly affecting gastrointestinal function or resection of the stomach or small bowel, symptomatic inflammatory bowel disease or ulcerative colitis, or partial or complete bowel obstruction.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2015-10-12 (Actual); Primary Completion 2019-11-15 (Actual); Study Completion 2020-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Margaret Tempero, MD, Principal Investigator — University of California, San Francisco
Locations (2):
- United States (2):
  - University of California, San Francisco, San Francisco, California
  - Oregon Health and Science University, Portland, Oregon

IPD SHARING:
Plan to Share IPD: Yes
Information from patient medical record may be shared with other participating institutions for safety monitoring.
Supporting Information: ICF

REFERENCES:
- [Derived] Sinha M, Betts C, Zhang L, Griffith MJ, Solman I, Chen B, Liu E, Tamaki W, Stultz J, Marquez J, Sivagnanam S, Cheung A, Pener D, Fahlman A, Taber E, Lerner K, Crocker M, Todd K, Rajagopalan B, Ware C, Bridge M, Vo J, Dragomanovich H, Sudduth-Klinger J, Vaccaro G, Lopez CD, Tempero M, Coussens LM, Fong L. Modulation of myeloid and T cells in vivo by Bruton's tyrosine kinase inhibitor ibrutinib in patients with metastatic pancreatic ductal adenocarcinoma. J Immunother Cancer. 2023 Jan;11(1):e005425. doi: 10.1136/jitc-2022-005425. PMID 36593070

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Dose Escalation for Safety and Toxicity | Immune Response Cohort
Started | 10 | 8
Completed | 10 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dose Escalation for Safety and Toxicity | Immune Response Cohort | Total
Number analyzed (Participants) | 10 | 8 | 18
Age, Customized [Count of Participants; unit: Participants]
  30-39 years | 0 | 1 | 1
  40-49 years | 1 | 0 | 1
  50-59 years | 4 | 1 | 5
  60-69 years | 3 | 4 | 7
  70-79 years | 1 | 1 | 2
  80-89 years | 1 | 1 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 4 | 10
  Male | 4 | 4 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 6 | 8 | 14
  Unknown or Not Reported | 3 | 0 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 0 | 0 | 0
  White | 4 | 7 | 11
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 5 | 0 | 5
Region of Enrollment [Number; unit: participants]
  United States | 10 | 8 | 18

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Who Experienced a Dose-Limiting Toxicity (DLT)
Description: DLTs will be based on the first course of treatment and defined as any unexpected grade 3 non-hematologic toxicity not reversible to grade 2 or less within 96 hours, or any grade 4 toxicity. Grade 4 hematological toxicities will not be considered dose limiting in this trial since a significant fraction of patients who are treated with gemcitabine and nab-paclitaxel are expected to experience these toxicities. Grade 3 peripheral neuropathy, a common and expected toxicity of treatment with nabpaclitaxel, will not be considered a DLT.
Time Frame: Up to 2 years
Measure: Number; unit: participants
Arm/Group | Dose Escalation for Safety and Toxicity | Immune Response Cohort
Number analyzed (Participants) | 10 | 8
participants | 9 | 8

2. Primary Outcome: Maximum Tolerated Dose (MTD)
Description: The dose level at which fewer than 2 of 6 patients experience a dose-limiting toxicity (DLT) will be designated as the Maximum Tolerated Dose (MTD)
Time Frame: Up to 2 years
Measure: Number; unit: mg/day
Arm/Group | Dose Escalation for Safety and Toxicity | Immune Response Cohort
Number analyzed (Participants) | 10 | 8
mg/day | 820 | 560

3. Primary Outcome: CA19-9 Clinical Response Rate
Description: The CA19-9 Response Rate is calculated using CA 19-9 treated patients who had a baseline CA19-9 > 75 units who have confirmed CA19-9 reduction of 75% from baseline value. Patients who have missing CA19-9 measurements will be treated as non-responders, i.e., they will be included in the denominator when calculating the percentage. The CA19-9 Response Rate, along with exact 95% confidence intervals, will be reported for the study.
Time Frame: 12 months
Population: Some patients did not have a decrease of 75% or did not have subsequent CA19-9 labs collected on study (i.e. off study prior to next time point) so they were not included in this analysis
Measure: Number (95% Confidence Interval); unit: proportion of responders
Arm/Group | Dose Escalation for Safety and Toxicity | Immune Response Cohort
Number analyzed (Participants) | 6 | 7
proportion of responders | 0.333 [0.0433 to 0.7772] | 0.143 [0.0036 to 0.5787]

4. Secondary Outcome: Median Time-to-progression (TTP)
Description: Time to Progression is defined as the time from date of first dose of protocol therapy to time of documented radiographic and/or clinical disease progression or death from any cause. Kaplan-Meier methods will be used to summarize median TTP with 95% confidence intervals.
Time Frame: 10 months
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Dose Escalation for Safety and Toxicity | Immune Response Cohort
Number analyzed (Participants) | 10 | 8
days | 128 [56 to NA] — The upper range of the confidence interval was calculated to be infinity | 126 [64 to NA] — The upper range of the confidence interval was calculated to be infinity

5. Secondary Outcome: Median Overall Survival (OS)
Description: Median OS for all enrolled patients will be calculated from date of first dose of protocol therapy until date of death, using chart review and/or follow up phone calls to determine date of death in patients after removal from study. The survival of patients still alive after 2 years of follow up post study discontinuation will be censored. Alive patients are censored at the date last known alive. Kaplan-Meier methods will be used to summarize median OS with 95% confidence intervals.
Time Frame: Up to 2 years
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Dose Escalation for Safety and Toxicity | Immune Response Cohort
Number analyzed (Participants) | 10 | 8
days | 246 [84 to NA] — The upper range of the confidence interval was calculated to be infinity | 170 [66 to NA] — The upper range of the confidence interval was calculated to be infinity

6. Secondary Outcome: Median Progression-free Survival (PFS)
Description: PFS is defined as the duration of time from date of first dose of protocol therapy to time of documented radiographic and/or clinical disease progression or death from any cause. Eligible patients are evaluable for PFS who are response-evaluable and who are removed from study for radiographic or clinical progression and/or who experience death from any cause during study follow up. Patients who have not progressed or died are censored at the date last known to be progression-free. Kaplan-Meier methods will be used to summarize median PFS with 95% confidence intervals. The proportion of patients with PFS equal to or exceeding 6 months will also be calculated and reported along with 95% confidence intervals.
Time Frame: 10 months
Measure: Median (Full Range); unit: days
Arm/Group | Dose Escalation for Safety and Toxicity | Immune Response Cohort
Number analyzed (Participants) | 10 | 8
days | 128 [56 to NA] — The upper range of the confidence interval was calculated to be infinity | 99 [64 to NA] — The upper range of the confidence interval was calculated to be infinity

ADVERSE EVENTS:
Time Frame: Up to 2 years
Arm/Group | Dose Escalation for Safety and Toxicity | Immune Response Cohort
All-Cause Mortality (participants affected / at risk) | 10/10 | 7/8
Serious Adverse Events (participants affected / at risk) | 5/10 | 3/8
Other Adverse Events (participants affected / at risk) | 10/10 | 6/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Escalation for Safety and Toxicity (N=10) | Immune Response Cohort (N=8)
Hepatobiliary disorders - Other (Hepatobiliary disorders) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Thromboembolic event (Vascular disorders) | 1 (1) | 0 (0)
Abdominal infection (Infections and infestations) | 0 (0) | 1 (1)
Infections and infestations - Other (Infections and infestations) | 0 (0) | 1 (2)
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
GI Bleed (Gastrointestinal disorders) | 1 (1) | 0 (0)
Blood Bilirubin increased (Investigations) | 2 (3) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Aspartate Aminotransferase (Investigations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Escalation for Safety and Toxicity (N=10) | Immune Response Cohort (N=8)
Nausea (Gastrointestinal disorders) | 7 (12) | 5 (12)
Diarrhea (Gastrointestinal disorders) | 5 (13) | 5 (8)
Vomiting (Gastrointestinal disorders) | 3 (4) | 3 (8)
Abdominal pain (Gastrointestinal disorders) | 5 (6) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 4 (4) | 0 (0)
Constipation (Gastrointestinal disorders) | 4 (5) | 0 (0)
Fatigue (General disorders) | 8 (17) | 3 (5)
Edema limbs (General disorders) | 7 (12) | 0 (0)
Fever (General disorders) | 3 (4) | 1 (1)
Platelet count decreased (Investigations) | 6 (17) | 2 (6)
Blood bilirubin increased (Investigations) | 2 (3) | 1 (1)
Weight loss (Investigations) | 2 (2) | 2 (2)
Neutrophil count decreased (Investigations) | 2 (3) | 1 (1)
Alkaline phosphatase increased (Investigations) | 2 (2) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 4 (6) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 4 (4)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 7 (7) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 4 (5) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (4) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 2 (3) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 7 (21) | 1 (2)
Dizziness (Nervous system disorders) | 4 (5) | 0 (0)
Dysgeusia (Nervous system disorders) | 2 (2) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 2 (4) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 4 (9) | 1 (1)
Depression (Psychiatric disorders) | 3 (3) | 0 (0)
Bloating (Gastrointestinal disorders) | 1 (1) | 1 (1)
Dry Mouth (Gastrointestinal disorders) | 2 (2) | 1 (1)
Gastritis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0)
Esophageal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 1 (1) | 0 (0)
Obstruction gastric (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oral hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Flu like symptoms (General disorders) | 1 (2) | 1 (1)
Edema Face (General disorders) | 1 (1) | 0 (0)
Facial Pain (General disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0)
Irritability (General disorders) | 1 (1) | 0 (0)
Thromboembolic event (Vascular disorders) | 2 (2) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Creatinine increased (Investigations) | 1 (1) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Nasal congestion (Reproductive system and breast disorders) | 2 (2) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 1 (1)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 (2) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1)
Lung infection (Infections and infestations) | 1 (1) | 0 (0)
Paronychia (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory infection (Infections and infestations) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 2 (2) | 0 (0)
Agitation (Psychiatric disorders) | 1 (1) | 0 (0)
Confusion (Psychiatric disorders) | 1 (2) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 2 (2)
Portal vein thrombosis (Hepatobiliary disorders) | 2 (2) | 1 (3)
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 2 (2) | 0 (0)
Bruising (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Cystitis noninfective (Renal and urinary disorders) | 1 (1) | 0 (0)
Hematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary tract pain (Renal and urinary disorders) | 1 (1) | 0 (0)
Allergic reaction (Immune system disorders) | 2 (2) | 0 (0)
Blurred Vision (Eye disorders) | 1 (1) | 0 (0)
Vaginal inflammation (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
Blood and lymphatic system disorders - Other (Blood and lymphatic system disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Treatment was determined to be ineffective and study was closed to accrual earlier than anticipated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2016-09-28): https://cdn.clinicaltrials.gov/large-docs/98/NCT02562898/Prot_SAP_001.pdf
  • Informed Consent Form (2018-04-24): https://cdn.clinicaltrials.gov/large-docs/98/NCT02562898/ICF_000.pdf